CLINICAL TRIAL: NCT05560646
Title: A Phase 2a/b, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter, Clinical Study to Evaluate the Efficacy and Safety of OG-6219 in 3 Dose Levels, in Women 18 to 49 Years of Age With Moderate to Severe Endometriosis-related Pain
Brief Title: A Study to Investigate Efficacy and Safety of OG-6219 BID in 3 Dose Levels Compared With Placebo in Participants Aged 18 to 49 With Moderate to Severe Endometriosis-related Pain
Acronym: ELENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OG-6219-P001
Record Dates: First submitted 2022-09-20; First posted 2022-09-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: Endometriosis Related Pain (ERP); Endometriosis; Pre-menopausal women
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: OG-6219 Dose 1 (Experimental): Group A: OG-6219 Dose 1 BID
  Interventions: Drug: OG-6219
- Group B: OG-6219 Dose 2 (Experimental): Group B: OG-6219 Dose 2 BID
  Interventions: Drug: OG-6219
- Group C: OG-6219 Dose 3 (Experimental): Group C: OG-6219 Dose 3 BID
  Interventions: Drug: OG-6219
- Group D: Placebo (Placebo Comparator): Group D: Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OG-6219 — OG-6219 Dose 1, Dose 2, Dose 3 BID: Participants will receive (orally) OG-6219 tablets during treatment cycles.
  Arms: Group A: OG-6219 Dose 1; Group B: OG-6219 Dose 2; Group C: OG-6219 Dose 3
Drug: Placebo — Participants will receive (orally) OG-6219 Placebo tablets BID during treatment cycles.
  Arms: Group D: Placebo

SUMMARY:
The purpose of this global Phase 2 study is to determine the efficacy, safety, and tolerability of 3 dose levels of OG-6219 in pre-menopausal women between 18 and 49 years of age (inclusive), who have moderate to severe endometriosis-related pain.

DETAILED DESCRIPTION:
This is a global multicenter, Phase 2a/b, randomized, double-blind, Placebo-controlled study to assess the efficacy, safety, and tolerability of 3 dose levels of OG-6219, in pre-menopausal women 18 to 49 years of age (inclusive), who have been surgically diagnosed with endometriosis with moderate to severe endometriosis-related pain. This study includes treatment lasting approximately 16 weeks in total and is followed by a Safety Follow-up visit.

Pre-menopausal females aged 18 to 49 years old (inclusive), who have been surgically diagnosed with endometriosis will be screened and randomly assigned to study treatment. A minimum subset of 10 participants per treatment group (including Placebo group) will be voluntarily enrolled for optional intensive PK sampling for the entire duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females of age 18 to 49 years old (inclusive) at the time of signing Informed Consent (V1).
* Surgically (laparoscopy or laparotomy) diagnosed with endometriosis
* Moderate to severe endometriosis-related pelvic pain
* Regular menstrual cycles
* Is not expected to undergo a planned gynecological surgery or other surgical procedures for treatment of endometriosis during study participation.
* Normal breast exam at V1. In participants of ≥40 years mammography or contrast-enhanced breast MRI performed within the last 12 months prior to Screening (V1) without clinically significant abnormal findings.
* Agree not to participate in another interventional study while participating in the present study.
* Able and willing to adhere to study procedures, including
* agree to use 2 forms of non-hormonal contraception throughout the study
* Must be willing and able to provide signed informed consent before any study-related activities
* Has demonstrated compliance with ≥75% of eDiary entries
* Has a negative pregnancy test

Exclusion Criteria:

* Surgical history of hysterectomy and/or bilateral oophorectomy
* Chronic pelvic and/or non-pelvic pain not caused by endometriosis that requires chronic analgesic or other chronic therapy
* Undiagnosed (unexplained), abnormal vaginal bleeding not associated with endometriosis within the past 6 months before screening.
* Presence of high-risk human papillomavirus (HPV).
* Has an active sexually transmitted infection (STI) (eg, gonorrhea, chlamydia, or trichomonas).
* Intends to become pregnant or breast feed during study participation or has a known or suspected pregnancy.
* History of malignancy (except for basal cell or squamous cell skin cancer) before signing informed consent.
* History of family history of hereditary abnormal hemoglobin or an enzyme deficiency that can result in methemoglobinemia.
* Has a medical condition associated with hemolytic anemia
* Known human immunodeficiency virus infection, and/or acute or active, recurrent/relapsing, or chronic infection (eg, hepatitis A, B, or C virus)
* Has a clinically significant abnormal ECG or QT interval prolongation
* Used any medication that is either a sensitive substrate, moderate, or strong inhibitor or inducer of CYP3A4 within 30 days or 10 half-lives (whichever is longer) prior to the planned first day of dosing.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Change from first treatment cycle to last planned treatment cycle in the mean OPP (endometriosis-related overall pelvic pain) score. The OPP measures endometriosis-related pain using NRS with range 0 (no pain) to 10 (worst imaginable). | First treatment cycle to last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
Safety and tolerability of OG-6219 | First treatment cycle through completion of follow-up, an average of 20 weeks (each cycle is approximately 28 days).
  Safety and tolerability of the treatment is assessed by proportion of participants who experienced any AEs/SAEs, abnormalities in clinical laboratory assessments, vital signs, and physical examination, and by proportion of participants who prematurely discontinued study treatment due to AEs/SAEs.

SECONDARY OUTCOMES:
Change from first treatment cycle to last planned treatment cycle in the mean DYS score | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
Change from first treatment cycle to last planned treatment cycle in the mean | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
  Non-menstrual pelvic pain (NMPP) scores. NMPP is a Numeric rating scale (NRS) that measures pain severity on a scale of 0 (no pain) to 10 (worst pain imaginable) where a lower value represents a better outcome.
Change from first treatment cycle to last planned treatment cycle in the mean dyspareunia score. | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
  Dyspareunia score is measured by the Endometriosis Pain Daily Diary on a numerical rating scale of 0-10 where 0=No Pain and 10=Worst Pain Imaginable. A lower value represents a better outcome.
Change from first treatment cycle to remaining treatment cycles in the mean number of tablets of rescue medication for endometriosis-related pain (ERP) and in the proportion of days participant has used rescue medication for ERP. | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
Change in Patient Global Impression of Severity (PGI-S) Score from V4 to Phone Contact 1, V6, and V7. | Visit 4 through V7, an average of 12 weeks (each cycle is approximately 28 days).
  The PGI-S is a 4-point response scale, over a 7-day recall period, measuring the overall severity of pelvic pain as: 0=none, 1=Mild, 2=Moderate, 3=Severe.
Percentage of participants with any improvement on the Patient Global Impression of Change at second, third and last planned treatment cycle. | Visit 4 through V7, an average of 12 weeks (each cycle is approximately 28 days).
Change from first treatment cycle to last planned treatment cycle in the Endometriosis Health Profile-30 (EHP-30) Domain Scores. | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days
  The EHP-30 consists of 30 items measured on a scale from 0 = Never to 4 = Always where the lower number represents a better outcome.
Mean change from Visit 1 to Visit 7 in bone biomarker levels | Screening through end of treatment, an average of 24 weeks.
Proportion of participants with clinical parameters of significance from Visit 1 to Visit 5, Visit 6, Visit 7, and Visit 8. | Screening through safety follow-up, an average of 28 weeks.
Mean change from first treatment cycle to second, third and fourth treatment cycles in the percentage of days with vaginal bleeding | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
ECG parameter changes at each of the four treatment cycle visits | First treatment cycle through completion of last planned treatment cycle, an average of 16 weeks (each cycle is approximately 28 days).
Mean change from V1 to V7 in serum hormone levels | Screening through end of treatment, an average of 24 weeks
Serum hormone levels at V5 comparing each treatment group | Visit 5
Serum hormone levels at V7 comparing each treatment group | At V7 approximately 24 weeks after patient consents to the study.
Plasma concentrations of OG-6219 and FOR-1011 at scheduled assessments using sparse PK sampling. | Second treatment cycle through completion of last planned treatment cycle, an average of 12 weeks (each cycle is approximately 28 days).
Cmax, for both OG-6219 and FOR-1011. | At 2 visits approximately 3 weeks apart beginning at second treatment cycle.
Tmax for both OG-6219 and FOR-1011 | At 2 visits approximately 3 weeks apart beginning at second treatment cycle
AucTAU for both OG-6219 and FOR-1011 | At 2 visits approximately 3 weeks apart beginning at second treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead Late-Stage Clinical Development, Study Director — Organon and Co
Locations (86):
- United States (27):
  - Central Research Associates LLC dba Flourish Research, Birmingham, Alabama
  - UAB Center for Women's Reproductive Health, Birmingham, Alabama
  - Olympia Clinical Trials, Los Angeles, California
  - Yale Fertility Center, Orange, Connecticut
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - MediSense Inc, Atlanta, Georgia
  - Paramount Research Solutions, College Park, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - The Advanced Gynecologic Surgery Institute, Park Ridge, Illinois
  - Ochsner Health Center - Baptist McFarland Medical Plaza, New Orleans, Louisiana
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - Bosque Women's Care, Albuquerque, New Mexico
  - University of Cincinnati, Cincinnati, Ohio
  - Centricity Research Dublin, Dublin, Ohio
  - Penn State Health Women's Health Clinic, Hershey, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Palmetto Clinical Research, Summerville, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Cedar Health Research, LLC, Euless, Texas
  - The Women's Hospital of Texas, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Tidewater Clinical Research, Norfolk, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Jan Palfijn Gent, Ghent
  - Universitair Ziekenhuis Ghent, Ghent
  - Jessa Ziekenhuis Hospital, Hasselt
  - CHU de Tivoli, La Louvière
- Bulgaria (10):
  - Medical Center Repromed EOOD, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - DCC " Ascendent" EAD, Sofia
  - SHATOD - Sofia District, EOOD, Sofia
  - MHAT for women's health - Nadezhda, OOD, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Group practice for specialized medical care in the field of obstetrics and gynecology - Gin Art OOD, Sofia
  - MHAT NiaMed OOD, Stara Zagora
  - Acibadem City Clinic MC Varna EOOD, Varna
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fertimed s.r.o., Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Femina Sana s.r.o., Prague
  - Ustav pro peci o matku a dite, Prague
- France (4):
  - Hopital Saint Joseph Paris, Paris, Paris
  - Hôpital Cochin, Paris
  - Hopital Tenon, Paris
  - Hospital of Hautepierre, Strasbourg
- Germany (3):
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Charité - Campus Benjamin Franklin, Berlin
  - Universitätsklinikum des Saarlandes, Homburg
- Hungary (5):
  - Clinexpert Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Anna Maganrendelo, Debrecen
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz, Nyíregyháza
- Italy (5):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Seriate, Milano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Roma
  - Università di Cagliari-Presidio Policlinico Monserrato, Monserrato
  - University of Siena Policlinico, Siena
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Latvia (3):
  - Latvian Maritime Medical Centre, Riga
  - Vitols & Vitols, Ltd., Riga
  - Dr. Vasaraudze's Private Clinic, Riga
- Poland (17):
  - Przychodnia Wielospecjalistyczna Sk-Medica Spółka Z O.O., Wroclaw, Dolnoslask
  - Specjalistyczna Poradnia Ginekologiczna Janusz Tomaszewski Spółka Komandytowa, Bialystok
  - Klinika Leczenia Niepłodności, Ginekologii i Położnictwa Bocian, Bialystok
  - Klinika Leczenia Niepłodności, Ginekologii i Położnictwa Bocian, Katowice
  - Clinical Medical Research Sp. z o.o., Katowice
  - NZOZ Medem, Katowice
  - Centra Medyczne Medyceusz, Lodz
  - Specjalistyczny Gabinet Ginekologiczno-Położniczy, Lublin
  - Centrum Medyczne Chodzki HLK, Lublin
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Etg Siedlce, Siedlce
  - Klinika Leczenia Niepłodności, Ginekologii i Położnictwa Bocian, Szczecin
  - MICS Centrum Medyczne Torun, Torun
  - Specjalistyczna Praktyka Lekar, Warsaw
  - PRATIA S.A. MTZ Clinical Research Powered by Pratia, Warsaw
  - WIM Panstwowy Instytut Badawczy Centralny Szpital Kliniczny MON, Warsaw
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Danderyd Sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.elenaendometriosisstudy.com/